CLINICAL TRIAL: NCT00964015
Title: Short-term Outcomes of Fluid Replacement and Resuscitation Strategy in the Cardiac Surgery Patient: A Randomized, Controlled Trial
Brief Title: Starch or Saline After Cardiac Surgery
Acronym: SSACS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of Funding
Sponsor: London Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Dave Nagpal, Associate Professor of Cardiac Surgery and Critical Care Medicine, Surgical Director of Heart Failure and Mechanical Circulatory Support Program, London Health Sciences Centre
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LHSC
Record Dates: First submitted 2009-08-20; First posted 2009-08-24 (Estimated); Last update posted 2019-08-15 (Actual); Status verified 2019-08

CONDITIONS: Coronary Artery Bypass Surgery
Keywords: colloid fluid; crystalloid fluid; surgery; coronary artery bypass grafting; renal function; Patients undergoing coronary artery bypass surgery
MeSH Terms: interventions — Hydroxyethyl Starch Derivatives; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Starch group (Active Comparator): Patients randomized to the Starch group will receive Voluven (6% Hydroxyethyl Starch 130/0.4) for their intravenous bolus and fluid resuscitation requirements.
  Interventions: Drug: 6% Hydroxyethyl Starch 130/0.4
- Saline group (Active Comparator): Patients randomized to the Saline group will receive 0.9% Normal Saline for their intravenous fluid bolus and resuscitation requirements
  Interventions: Drug: 0.9% Normal Saline

INTERVENTIONS:
Drug: 6% Hydroxyethyl Starch 130/0.4
  Arms: Starch group
Drug: 0.9% Normal Saline
  Arms: Saline group

SUMMARY:
When people undergo major surgery, they require intravenous supplementation of fluids for a number of reasons:

* to compensate for no oral intake
* to support blood pressure and organ function during and after surgery
* to replace lost fluid or blood volume

There are a variety of fluid choices doctors have to provide to patients, and it is still not definitively known whether some fluids are better than others in specific situations. This is a particularly interesting question in patients undergoing heart surgery because of the significant volume of fluids used over the entire course of hospitalization, including before the operation, during the operation, and after the operation.

There has been some scientific evidence that the use of starch-based fluids (synthetic colloids) leads to better oxygen delivery to the organs with a smaller volume of fluid given, providing for better recovery from surgery. However, there has also been some scientific evidence that the use of these fluids can harm kidney function. Importantly, none of these large-scale studies were carried out specifically in patients undergoing heart surgery.

The purpose of this study is to answer the question of whether the use of starch-based fluid in the heart surgery patient makes for a safer and faster recovery, causes kidney dysfunction, or makes no discernable difference.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing elective primary isolated on-pump coronary artery bypass grafting

Exclusion Criteria:

* pregnant patients
* patients with an active intra-cranial bleed
* patients with a history of hypersensitivity to starch solutions
* patients with Stage 4 or 5 Kidney Disease (estimated glomerular filtration rate < 30 ml / min / 1.73 m2)
* patients with a significant preoperative metabolic acidosis, defined by a preoperative capillary blood pH less than or equal to 7.2 and a serum bicarbonate less than 15

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2009-08 (Actual); Primary Completion 2010-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Incidence of acute kidney injury as defined by RIFLE criteria | Short term (in hospital, up to 30 days) and mid-term (2 months)
Maximum postoperative weight gain | Short-term (in hospital, up to 7 days)

SECONDARY OUTCOMES:
Operative mortality | In hospital (up to 30 days)
Duration of ventilation support requirements | In hospital (up to 30 days)
Total chest tube drainage (until removed) | In hospital (up to 30 days)
ICU length of stay | In hospital (up to 30 days)
Transfusion of blood products | In hospital (up to 30 days)
Incidence of atrial fibrillation (necessitating a change in medical management) | In hospital (up to 30 days)
Duration of oxygen supplementation | In hospital (up to 30 days)
Creatinine, Urea, Cr Clearance as estimated by the MDRD formula | In hospital at defined timepoints, and at 2 months post hospital discharge
Volume of fluid infused | In hospital (up to 7 days)
Total hospital length of stay (when ready to leave tertiary hospital setting) | In hospital

CONTACTS AND LOCATIONS:
Overall Officials: Dave Nagpal, MD, Study Director — LHSC / UWO; Ray Guo, MD, Principal Investigator — LHSC / UWO; Chris Harle, MD, Principal Investigator — LHSC / UWO
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada